CLINICAL TRIAL: NCT02298855
Title: A Randomised Study Comparing Satisfaction With Individualised Follow-up Led by a Trained Cancer Nurse Versus Conventional Medical Follow-up After Primary Treatment for Ovarian Cancer.
Brief Title: Individualised Versus Conventional Medical Follow-up for Women After Primary Treatment for Ovarian Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other); Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OC_F-UP_V3 28/07/2006
Record Dates: First submitted 2014-09-30; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-09

CONDITIONS: Ovarian Cancer
Keywords: Gynaecological cancer; Nurse-led care; Aftercare; Patient self-management; Quality of life; Relapse free interval; Watch and wait
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional follow-up (No Intervention): Treatment as usual will involve: one post treatment appointment then 3 monthly appointments with a Dr. At appointments: medical history; investigations to monitor disease progression including CA125 tumour marker blood test if this were raised at diagnosis. A physical examination may be performed.
- Individualised follow-up (Experimental): Follow-up is delivered by a nurse and frequency and type (telephone or face-to-face) is negotiated to suit their individual situation. Assessment by holistic guide. The intervention is informed by a model of health promoting interactions oriented towards improving self-efficacy. The nurses will provide information and support to help patients manage symptoms and psychological discomfort.
  Interventions: Behavioral: Individualised follow-up

INTERVENTIONS:
Behavioral: Individualised follow-up — Patients allocated to gynaecological cancer nurse specialist at the end of primary treatment. Follow-up is negotiated to suit their individual situation. Type of contact is flexible, primarily by telephone although some women may opt for face-to-face appointments. Patients will be assessed using a holistic guide to identify signs of disease progression, symptoms warranting intervention, and psychological issues. The nurses delivering the intervention are expert in the management of ovarian cancer and will work to a model of health promoting interactions oriented towards improving self-efficacy. The nurses will provide information and support to assist patients to manage troublesome symptoms and live with psychological discomfort.
  Arms: Individualised follow-up

SUMMARY:
The purpose of this study in women who have completed primary treatment for ovarian cancer is to investigate the effects of individualised follow-up care delivered by a nurse compared to conventional medical follow-up on quality of life and mood. The investigators aim to determine if the individualised treatment is acceptable to women compared to the conventional treatment.

DETAILED DESCRIPTION:
There is recent evidence that routine cancer follow-up is ineffective (Kew, 2011). Knowledge of how best to deliver follow-up remains inadequate and randomised studies are lacking. This trial compares individualised follow-up led by a cancer trained nurse to conventional medical follow-up.

Aim:

The investigators shall conduct the trial using experienced clinical nurse specialists (CNSs) to deliver self-management focused individual follow-up and evaluate whether this brings about greater improvement in quality of life, is acceptable and cost saving when compared to the standard (conventional) model.

Design:

Two arm randomised controlled trial.

Setting:

Specialist gynaecological cancer outpatient services at three cancer centres, one inner city and two urban.

Sample size:

A sample size of 100 patients, randomised equally to the 2 treatment groups, has been determined for this study. See statistical analysis section.

Recruitment:

Based on previous experience of recruiting in this population approximately 50% of women approached will agree to take part. The investigators need 1 year to recruit the sample.

Randomisation:

Participants will be subdivided into two groups those recruited at the inner city centre and those recruited at the suburban. Randomisation will be performed independently for both groups with participants randomly allocated to either the conventional or individualised follow-up in a 1:1 ratio. Allocation of the first participant from a pair to one of the 2 follow-up strategies will be made using randomness derived from atmospheric noise (http://www.random.org); the second participant from each pair will then be allocated to the other group.

The intervention:

Trial follow-up is 2 years from baseline. Conventional follow-up/treatment as usual This will remain unchanged and involve: one post treatment appointment then appointments every 3 months with a doctor. Routinely a medical history is taken and investigations to monitor disease progression including serum cancer antigen 125 (CA125) tumour marker. A physical examination may be performed. The appointment will sometimes involve CNS input and patients may contact the non-study CNS on an ad hoc basis.

Individualised follow-up Patients will meet the study CNS in clinic when they attend for their 4-6 week post treatment appointment. The nurse will negotiate with the patient to agree follow-up arrangements best suited to their needs. E.g. patient-initiated telephone or face-to-face appointments. The nurse will assess the patient at appointments using an assessment proforma.

Data collection:

Quantitative data Baseline qol questionnaires will be provided by the Research Assistant at the time of written consent and completed and returned prior to disclosure of randomisation. Subsequent questionnaires will be posted to participants with a reply paid envelope.

Data will be entered on a 'Patient events' data base and then extracted for all patients for different types of service use during the two-year follow-up period. The investigators will also record primary care contacts and the reasons for these with a questionnaire to General Practitioners.

Qualitative interview data Selected patients will take part in a 45-60 minute one-to-one interview at a location convenient to them. The interview will be audio-recorded following consent and anonymised to maintain confidentiality. A semi-structured interview guide will be used to ensure all important topic areas are covered.

CNSs will be interviewed in a quiet room away from their clinical area as above.

Data Analysis:

Quantitative data Differences in mean patient qol and satisfaction and between the two groups will be assessed by 2 sample t-tests. Assuming a two-sided significance level of 5% with 40 in each sample, to achieve 80% power any differences will have to be quite large to be detectable. For the satisfaction scale (0-100), where the estimated common standard deviation = 14.7 (de Bock et al (2004)), a difference between the two groups of 9.3 would be detectable with 80% power. For the anxiety (0-13) and depression (0-14) measures common standard deviation = 2.75 in both cases (de Bock et al 2004), such a difference would need to be 1.74 in both cases. The investigators may be able to detect smaller differences with the planned sample size when taking into account adjustment for baseline values in the sample size calculation comparing the randomised groups (analysis of covariance).

For the qol scales there are various sub-scales (0-100) and the evidence from literature sources suggest that for most scales the standard deviation is approximately 20-25 (Greimel et al 2003). Using such a value then, a difference in means, detectable with 80% power, would be between 12.7 and 15.9. Even if the ensuing results are not able to detect clinically important differences between the two groups, the scale scores will provide useful information and may justify further inquiry.

The total cost of follow-up for each patient will be calculated by multiplying service use by unit costs obtained from relevant National Health Service (NHS) Reference Costs and summing across all types of use. Unadjusted service use and total costs will be compared between each group using Mann-Whitney two-sample statistics.

Qualitative data Interviews will be fully transcribed and analysed according to principles of grounded theory (Strauss and Corbin, 1991).

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of ovarian cancer (includes fallopian tube and peritoneal cancers)
2. Within one month of completion of primary treatment including surgery & chemotherapy/radiotherapy or surgery alone, irrespective of outcome with regard to remission
3. Expected survival ≥3 months
4. Agreement to be randomised
5. Agreement to give written consent to participate in the study
6. Sufficient grasp of English to engage in the self-management focused approach.

Exclusion Criteria

1. A second cancer diagnosis
2. Clinician estimated survival of ≤ 3 months
3. Women receiving treatment for a mental health condition
4. Women who have a learning disability.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-01; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The European Organisation for Research and Treatment of Cancer (EORTC) core quality of life questionnaire QLQ-C30 with ovarian cancer specific module Ov-28. | Assessment of change over time from baseline and at 3, 6, 12,18, & 24 months.
  is a 30-item questionnaire assessing five 5 functional domains (physical, role, cognitive, emotional and social), 3 symptom domains (nausea/vomiting, fatigue and pain), and a number of specific symptoms (dyspnoea, appetite loss, sleep disturbance, constipation, and diarrhoea) as well as the perceived financial impact of the disease and treatment.The site specific instrument (Ov-28) used with the QLQ-C30 consists of 28 items which are factor analysed into six factors: abdominal/gastrointestinal symptoms, peripheral neuropathy, other chemotherapy side effects specific to ovarian cancer treatments, hormonal symptoms, body image and sexuality, and attitude to disease/treatment. Higher scores for functioning subscales indicate better functioning. Higher scores in symptom subscales indicate worse symptoms.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS): | Assessment of change over time from baseline and at 3, 6, 12, 18, & 24 months.
  Hospital Anxiety and Depression Scale (HADS): Anxiety and depressive symptoms will be assessed with this 14-item self-rated scale designed for use in the medically ill.

OTHER OUTCOMES:
Ware Patient Satisfaction Questionnaire (PSQ-III) to measure patients' perceptions of care. | Asssessment of change over time from baseline and at 3, 6, 12, 18, and 24 months.
  This provides a summary measure, general satisfaction, as well as six aspects of health care: technical competence, interpersonal manner, communication, time spent with clinician, financial aspects, and access to care. In the version we will use the financial items will be left out because these are not appropriate for the UK national socialised health system.
Qualitative interviews with 20-24 selected patients receiving conventional or individualised follow-up care. | Between 1 & 2 years on follow-up.
  Findings from the questionnaires at 6 and 18 months will be used to purposively select a sub-sample of 10-12 women from each arm of the study for in-depth interview. Women will be selected to maximise variation in terms of quality of life scores, patient satisfaction and HADS scores in each arm of the study. Care will also be taken to include women of different ages and ovarian cancer stage. Patients' experiences of follow-up and their preferences for follow-up care will be elicited in one-to-one semi-structured interviews which will be conducted by the clinical psychologist, a co-investigator to the project.
Qualitative interviews with 4 clinical nurse specialists delivering the intervention | After 1 & 2 years and during delivery follow-up care to study participants.
  Nurses' experiences of delivering the follow-up care will be elicited in one-to-one semi-structured interviews to be conducted by the clinical psychologist, a co-researcher to the project.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lanceley, PhD, Principal Investigator — University College, London
Locations (3):
- United Kingdom (3):
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, Essex.
  - Basildon & Thurrock University Hospitals NHS Foundation Trust, Basildon, Essex
  - University College London Hospital NHS Foundation Trust, London, London

REFERENCES:
- [Background] Greimel E, Bottomley A, Cull A, Waldenstrom AC, Arraras J, Chauvenet L, Holzner B, Kuljanic K, Lebrec J, D'haese S; EORTC Quality of Life Group and the Quality of Life Unit. An international field study of the reliability and validity of a disease-specific questionnaire module (the QLQ-OV28) in assessing the quality of life of patients with ovarian cancer. Eur J Cancer. 2003 Jul;39(10):1402-8. doi: 10.1016/s0959-8049(03)00307-1. PMID 12826043
- [Background] Kew F, Galaal K, Bryant A, Naik R. Evaluation of follow-up strategies for patients with epithelial ovarian cancer following completion of primary treatment. Cochrane Database Syst Rev. 2011 Jun 15;(6):CD006119. doi: 10.1002/14651858.CD006119.pub2. PMID 21678351
- [Background] de Bock GH, Bonnema J, van der Hage J, Kievit J, van de Velde CJ. Effectiveness of routine visits and routine tests in detecting isolated locoregional recurrences after treatment for early-stage invasive breast cancer: a meta-analysis and systematic review. J Clin Oncol. 2004 Oct 1;22(19):4010-8. doi: 10.1200/JCO.2004.06.080. PMID 15459225